CLINICAL TRIAL: NCT05762289
Title: A Randomized Control Trial Comparing the Immediate Effects Cervical Thrust Manipulation in Weight Bearing and Non Weight Bearing Position for Improving Cervical Range of Motion and Pain in Forward Head Posture
Brief Title: Comparison of Weight Bearing Thrust Manipulation With Non Weightbearing Thrust Manipulation in Patients With Forward Head Posture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yusra Medical and Dental College (Other)
Responsible Party: Principal Investigator, Maham Nasir, Head Of Physical Therapy Department, Yusra Medical and Dental College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YusraMDC
Record Dates: First submitted 2023-02-23; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Cervical Pain
Keywords: forward head posture, cervical thrust manipulation
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Masking Description: Patients were randomized using sealed envelope method where all the participants selected their envelopes which were opaque and placed in a container . All the patients who were willing after informing all the risk and procedures were then selected in two groups Group A (treatment group) or weight bearing group and Group B (Control group)non weight bearing group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Change in range of motion and within the weight bearing group (Experimental): . Subjects in Group A or treatment group were seated and given thrust manipulation using belt. Cervical spine was placed in neutral position and belt was stabilized on C4-C5 which is the part that causes most stiffness and pain and lost of range. Patient placed belt in left hand for left sided thrust and caudal force was applied , therapist held other end of the belt and applied stretch in the line of eye ball. The cervical spine of patient was guided in left rotation until resistance was felt and than thrust of high velocity low amplitude was given by therapist . This was done for both sides if the cavitation sound was not heard manipulation was tried for a second time after 10 minutes by repositioning the patient but no more than two times in a day. Therapist performing manipulation was skilled in giving belt thrust manipulation.
  Interventions: Other: Thrust Manipulation (in weight bearing and non weight bearing)
- Control (Active Comparator): While Group B received manipulation in supine position by maitland's traditional thrust. Where the neck is slightly flexed by therapist hand on the occipit where therapist is standing behind the head. Neck is guided in right side flexion and opposite rotation and at the end of rang high velocity low amplitude thrust is applied. This was done for both sides if the cavitation sound was not heard manipulation was tried for a second time after 10 minutes by repositioning the patient but no more than two times in a day
  Interventions: Other: Thrust Manipulation (in weight bearing and non weight bearing)

INTERVENTIONS:
Other: Thrust Manipulation (in weight bearing and non weight bearing) — Pain and Range of cervical motion was assessed before and after manipulation in both groups.

SUMMARY:
This randomized controlled trial was performed in MMRC (Majestic medicine rehabilitation Sciences) Islamabad in February 2023 and consisted of patients having neck pain and forward head posture. 30 Patients were divided into two groups of 15 each by sealed envelope method . Treatment group was given weight bearing thrust manipulation in sitting and control was given non weight bearing thrust manipulation in supine lying. Pain was calculated through NPRS and Cervical ranges were calculated by Inclinometer before and immediately after treatment.

DETAILED DESCRIPTION:
Cervical Spine is most integral part of human spine as it sits between highly stable thoracic and highly movable occipital bodies. It help the head movement of flexion , rotation which are constantly required for performing basic activities of daily life. It is a link between head and rest of the body and due to its need in mobility it is often put under greater stress , muscular imbalance, reduced disc spaces and common site for many spinous syndromes. One of the most common disability that occurs on cervical spine is forward headv posture usually associated with upper crossed syndrome and is known as text neck also due to strain put on spine due to high usage of screen devices. Sedentary lifestyle and postural imbalances and effect of gravity are usually the major causes of muscular and bony imbalances that result in forward head posture. Prolonged state of stress on muscles usually result in pain in neck specially during movement.

High Velocity Low Amplitude Thrust (HVLAT) is a common technique to unlock cervical joints and muscular pain associated with it and immediately reduce pain. Cavitation sound or pop is often associated with this thrust technique that is result decrease in pressure causes dissolved gasses in the synovial fluid to be released into the joint cavity of due to which , the force-displacement curve shifts and the range of motion of the joint increases.It has been stated that spinal manipulation activates presynaptic inhibition of segmental pain pathways, reflex muscle relaxation, and reflex pain Inhibition. It has been repeatedly proved by literature that thrust manupulation is an effective was of increasing ROM and pain in patients in non weight bearing positions but it can also be given in weight bearing position effects of which are yet not very clear specially in patient population such as forward head posture .The current study was planned to compare the effectiveness of thrust manipulation in weight bearing and non weight bearing postions on pain and range in forward head posture . The hypothesis was that there will be significant difference in the effect of thrust manipulation in different positions.

ELIGIBILITY:
Inclusion Criteria

* Forward head posture
* Patients who had complain of neck pain
* Decrease range of flexion, extension, rotation and side flexion of cervical spine
* Craniovertebral angle below 48 were included

Exclusion Criteria :

* Patients with structural or anatomical deformity,
* recent surgical history , degenerative changes ,
* cervical instability,
* malignancy
* radiculopathy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Change in Neck pain before and after thrust manipulation | As immediate effects are measured pain before giving manipulation and 10minutes after session is measured
  pain will be calculated using Numeric pain rating scale(NPRS) before and after manipulation
Change in Cervical Range of motion before and after thrust manipulation | As immediate effects are measured ranges of motion before giving manipulation and 10minutes after session is meas
  Range Of Motion will be measured using inclinometer before and after manipulation

CONTACTS AND LOCATIONS:
Overall Officials: Maham Nasir, DPT, Principal Investigator — Yusra institute of Rehabilitation sciences
Locations (1):
- MMRC, Islamabad, Pakistan